CLINICAL TRIAL: NCT04890834
Title: Improving Healthcare Utilization and Quality of Life in Head and Neck Cancer Patients Undergoing Chemoradiation and Their Family Caregivers
Brief Title: Dyadic Yoga Intervention for the Improvement of Healthcare Utilization and Quality of Life in Patients With Head and Neck Cancer Undergoing Chemoradiation and Their Caregivers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0311; NCI-2020-13884 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0311 (Other: M D Anderson Cancer Center); R01CA247307 (NIH)
Record Dates: First submitted 2021-01-27; First posted 2021-05-18 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Standard of care) (Active Comparator): Patients and caregivers receive standard care including education pertaining to symptom management, prophylactic dental hygiene and possible extraction, speech pathology for baseline swallowing assessment and prophylactic treatment, and dietary services for regular nutrition consults during CRT. Psychiatry, social work, interventional radiology and supportive care services are consulted as needed.
  Interventions: Other: Best Practice; Other: Questionnaire Administration
- Arm II (exercise, yoga sessions) (Other): Patients and caregivers receive standard care as in arm I. Patients and caregivers also participate in yoga sessions 3 times per week over 60 minutes each for a total of 15 sessions.
  Interventions: Other: Best Practice; Other: Exercise Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard care
  Other Names: standard of care; standard therapy
Other: Exercise Intervention — Participate in yoga sessions
  Arms: Arm II (exercise, yoga sessions)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This study evaluates if partner-based (dyadic) yoga programs may improve the quality of life of patients with head and neck cancer undergoing chemoradiation and their caregivers, and if it is a cost-effective option. Yoga programs may decrease how often patients come to the hospital during and after treatment with chemoradiation, and improve the quality of life for both patients and caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the efficacy of the dyadic yoga (DY) intervention regarding reduced patient emergency department (ED) visits and feeding tube (FT) insertions and improved patient and caregiver quality of life (QOL) as compared to the usual care (UC) group.

II. Estimate intervention costs, direct medical costs, indirect costs (i.e., productivity loss), and evaluate the overall cost-effectiveness of the DY intervention for patients and caregivers.

III. Demonstrate that, compared to the UC group, the DY program improves patient and caregiver symptoms burden, objective physical function, and illness communication and reduces patient use of opioids during chemoradiotherapy (CRT), which will in turn mediate intervention outcomes at the follow-up assessments.

IV. Understand the patient and caregiver experience of head and neck cancer (HNC), healthcare utilization and symptom management and emerging themes as possible mediators as they relate to or suggest modifications of our proposed model using qualitative methods.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Patients and caregivers receive standard care including education pertaining to symptom management, prophylactic dental hygiene and possible extraction, speech pathology for baseline swallowing assessment and prophylactic treatment, and dietary services for regular nutrition consults during CRT. Psychiatry, social work, interventional radiology and supportive care services are consulted as needed.

ARM II: Patients and caregivers receive standard care as in arm I. Patients and caregivers also participate in yoga sessions 3 times per week over 60 minutes each for a total of 15 sessions.

After completion of study, participants are followed up every 2 weeks for 3 months and then monthly for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Diagnosed with a primary HNC and going to receive at least 5 weeks (25 fractions) of CRT
* PATIENTS: Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* PATIENTS: Having a family caregiver (e.g., spouse/partner, sibling, adult child) willing to participate
* PATIENTS AND CAREGIVERS: Must be at least 18 years old
* PATIENTS AND CAREGIVERS: Able to read and speak English
* PATIENTS AND CAREGIVERS: Able to provide informed consent

Exclusion Criteria:

* PATIENTS AND CAREGIVERS: Who have regularly (self-defined) participated in a yoga program in the year prior to diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient healthcare utilization (Standard of care) | Up to 6 months with 3 months follow-up
  Will examine group differences in patient emergency department visit (yes/no) during the observation period of during and up to 3 months post chemoradiotherapy (CRT) as the primary outcome. Will use logistic regression with the randomization factors as covariates, as these factors may be associated with the study outcomes, and controlling for them is likely to increase the power to detect the between-group differences.

SECONDARY OUTCOMES:
Caregiver quality of life questionnaire (RAND 36-Item Health Survey) | Up to 6 months with 3 months follow-up
  Will examine group differences over the 6-month follow-up period specifying the T4 as the primary endpoint using a dyadic model (assuming additional dependence in outcomes between patient and caregiver outcomes). This analysis will be imbedded in a linear mixed-effects (alternatively known as the multilevel) model analysis, with repeated measures over time (i.e., at end of CRT, 1-, 3- and 6-month follow-ups). In the mixed models, group will be entered as a primary variable of interest and baseline level of the outcome will be treated as a covariate.
  Participants Energy/Fatigue level-(0-lowest energy level/ 100-highest energy no fatigue)
Patient quality of life questionnaire | Up to 6 months with 3 months follow-up
  Will examine group differences over the 6-month follow-up period specifying the T4 as the primary endpoint using a dyadic model (assuming additional dependence in outcomes between patient and caregiver outcomes). This analysis will be imbedded in a linear mixed-effects (alternatively known as the multilevel) model analysis, with repeated measures over time (i.e., at end of CRT, 1-, 3- and 6-month follow-ups). In the mixed models, group will be entered as a primary variable of interest and baseline level of the outcome will be treated as a covariate.
  Participants Energy/Fatigue level-(0-lowest energy level/ 100-highest energy no fatigue)

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org